CLINICAL TRIAL: NCT04957784
Title: Study on the Current Situation and Related Factors of Hypertension Management in a Poor County in Shanxi Province
Status: Completed | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: LM2021110
Record Dates: First submitted 2021-06-29; First posted 2021-07-12 (Actual); Last update posted 2021-07-12 (Actual); Status verified 2021-06

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: questionnaire survey — Understand the current situation of hypertension management in a poor county in Shanxi Province through questionnaire surveys, and explore the factors that affect patients' blood pressure control based on local conditions

SUMMARY:
This project aims to understand the current situation of hypertension management in a poor county in Shanxi Province, and explore the factors that affect patients' blood pressure control based on local reality, and provide a basis for further promoting the standardized management of hypertension in poor areas and the comprehensive prevention and control of chronic diseases at the national grassroots level.

ELIGIBILITY:
Inclusion Criteria:

（1）Clinical diagnosis of hypertension (2) Permanent population or floating population who have lived for more than 6 months in the area; (3) In the case of not taking antihypertensive drugs, after 3 different daily blood pressure measurements, the systolic blood pressure ≥140 mmHg and/or the diastolic blood pressure ≥90 mmHg were achieved in all 3 times, and it has been diagnosed by the community and above medical institutions in the past. Residents with high blood pressure; (4) As of October 2020, all research subjects have been included in the national basic public health service projects by medical institutions and have received standardized management of hypertension for one full year.

Exclusion Criteria:

1. Pregnant and lactating women;
2. Those who are critically ill, mentally ill, cognitively impaired, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hypertensive population in a poverty-stricken county of Shanxi Province
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-05-30 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
questionnaire survey | 6 months
  General demographic characteristics, lifestyle, medication status, health knowledge awareness

CONTACTS AND LOCATIONS:
Overall Officials: Gaiqi Yao, Study Chair — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, China